CLINICAL TRIAL: NCT00420316
Title: To Assess Long-term Efficacy & Safety of Subjects Approximately 3 Years After Priming With 2 Doses of GlaxoSmithKline (GSK) Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine (Rotarix) in the Primary Vaccination Study (102247).
Brief Title: Long-term Efficacy and Safety of Subjects Approximately 3 Years After Priming With 2 Doses of GSK Bio's HRV Vaccine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109810
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Infections, Rotavirus
Keywords: Intussusception; Gastroenteritis; Finland
MeSH Terms: conditions — Rotavirus Infections; Intussusception; Gastroenteritis | interventions — RIX4414 vaccine

ARMS (2):
- Rotarix Group (Experimental): Healthy children between and including 6 to 12 weeks of age at the time of first vaccination, who received two powdered oral doses of Rotarix™ vaccine in the Rota-036 primary vaccination study (102247), were subsequently followed-up for 6 months during their third year of age, in scope of the present study.
  Interventions: Biological: Rotarix (primary vaccination study)
- Placebo Group (Placebo Comparator): Healthy children between and including 6 to 12 weeks of age at the time of first vaccination, who received two liquid oral doses of placebo in the Rota-036 primary vaccination study (102247), were subsequently followed-up for 6 months during their third year of age, in scope of the present study.
  Interventions: Biological: Placebo (primary vaccination study)

INTERVENTIONS:
Biological: Rotarix (primary vaccination study) — GlaxoSmithKline Biologicals' oral live attenuated human rotavirus vaccine.
  Arms: Rotarix Group
Biological: Placebo (primary vaccination study) — Two liquid oral doses of placebo
  Arms: Placebo Group

SUMMARY:
To assess the long-term efficacy and safety of the subjects during the third year after priming with 2 doses of GSK Biologicals' oral live attenuated HRV vaccine (Rotarix) in the primary vaccination study (102247). The Rotarix vaccine was administered in the primary vaccination study. There was no vaccine/intervention in this long-term efficacy study.

ELIGIBILITY:
Inclusion Criteria:

* A male or female who has completed the second year efficacy follow-up of the primary vaccination study in Finland.
* Written informed consent obtained from the parent or guardian of the subject.

Ages: 32 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1613 (Actual)
Dates: Start 2007-02-12 (Actual); Primary Completion 2007-08-08 (Actual); Study Completion 2007-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Finland (12):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 109810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Rotarix Group | Placebo Group
Started | 1082 | 531
Completed | 1070 | 522
Not Completed | 12 | 9
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix Group | Placebo Group | Total
Number analyzed (Participants) | 1082 | 531 | 1613
Age, Continuous [Mean (Standard Deviation); unit: Months] | 31.2 (1.12) | 31.3 (1.19) | 31.23 (1.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 510 | 266 | 776
  Male | 572 | 265 | 837

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Rotavirus Gastroenteritis (RVGE)
Description: Occurence of any rotavirus gastroenteritis (RVGE) caused by the circulating wild-type rotavirus strain was assessed in terms of number of subjects experiencing diarrhoea with or without vomiting. Two occurrences of diarrhoea were classified as separate episodes if there were 5 or more diarrhoea-free days between the episodes.
Time Frame: During the study period for the long-term follow-up (i.e. 6 months)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, which included all subjects from the ATP efficacy cohort of the primary study (102247) who entered into the efficacy surveillance period.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1065 | 525
Subjects | 4 | 3
Statistical Analysis 1: Comparison: Rotarix Group vs Placebo Group; Vaccine efficacy with respect to any rotavirus gastroenteritis (RV GE) caused by the circulating wild-type rotavirus strain. Vaccine efficacy (VE) was defined as the percent reduction in the frequency of the relevant outcome variable in vaccinated subjects compared with those subjects who received placebo; Test type: Superiority or Other; p = 0.691, Fisher Exact; Percent reduction = 34.3, 95% CI 2-sided [-348.7 to 88.9]

2. Secondary Outcome: Number of Subjects With Severe Rotavirus Gastroenteritis (RVGE)
Description: Number of rotavirus gastroenteritis (RVGE) episodes caused by the wild-type rotavirus strain and reported during the efficacy period, were presented by severity, using the Vesikari scale. The assessment of intensity of GE episodes was done using the 20-point Vesikari scale, according to which episodes with scores greater than or equal to (≥) 11 were labeled as severe.
Time Frame: During the study period for the long-term follow-up (i.e. 6 months)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1065 | 525
Subjects | 1 | 1
Statistical Analysis 1: Comparison: Rotarix Group vs Placebo Group; Vaccine efficacy with respect to severe rotavirus gastroenteritis (RVGE) caused by the circulating wild-type rotavirus strain was assessed. Vaccine efficacy (VE) was defined as the percent reduction in the frequency of the relevant outcome variable in vaccinated subjects compared with those subjects who have received placebo; Test type: Superiority or Other; p = 0.551, Fisher Exact; Percent reduction = 50.7, 95% CI 2-sided [-3769.6 to 99.4]

3. Secondary Outcome: Number of Subjects With Any Rotavirus Gastroenteritis (RVGE) With G1 Serotype
Description: Occurence of any rotavirus gastroenteritis (RVGE) caused by the circulating wild-type rotavirus strain was assessed in terms of number of subjects experiencing diarrhoea with or without vomiting. Two occurrences of diarrhoea were classified as separate episodes if there were 5 or more diarrhoea-free days between the episodes. Only GE episodes in which wild-type RV strain of G1 serotype was identified in a stool specimen, were included in the efficacy analysis.
Time Frame: During the study period for the long-term follow-up (i.e. 6 months)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1065 | 525
Subjects | 0 | 2

4. Secondary Outcome: Number of Subjects With Severe Rotavirus Gastroenteritis (RVGE) With G1 Serotype
Description: Number of rotavirus gastroenteritis (RVGE) episodes caused by the wild-type rotavirus strain of serotype G1 and reported during the efficacy period, were presented by severity, using the Vesikari scale. The assessment of intensity of GE episodes was done using the 20-point Vesikari scale, according to which episodes with scores greater than or equal to (≥) 11 were labeled as severe.
Time Frame: During the study period for the long-term follow-up (i.e. 6 months)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1065 | 525
Subjects | 0 | 1
Statistical Analysis 1: Comparison: Rotarix Group vs Placebo Group; Vaccine efficacy with respect to severe rotavirus gastroenteritis (RVGE) caused by the wild-type rotavirus strain of serotype G1. Vaccine efficacy (VE) was defined as the percent reduction in the frequency of the relevant outcome variable in vaccinated subjects compared with those subjects who received placebo; Test type: Superiority or Other; p = 0.33, Fisher Exact; Percent reduction = 100, 95% CI 2-sided [-1822.5 to 100]

5. Secondary Outcome: Number of Subjects With Any Rotavirus Gastroenteritis (RVGE) With Non-G1 Serotype
Description: Occurence of any rotavirus gastroenteritis (RVGE) caused by the circulating wild-type rotavirus strain of non-G1 serotype was assessed in terms of number of subjects experiencing diarrhoea with or without vomiting. Two occurrences of diarrhoea were classified as separate episodes if there were 5 or more diarrhoea-free days between the episodes.
Time Frame: During the study period for the long-term follow-up (i.e. 6 months)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1065 | 525
Subjects | 4 | 1
Statistical Analysis 1: Comparison: Rotarix Group vs Placebo Group; Vaccine efficacy with respect to any rotavirus gastroenteritis (RVGE) caused by the wild-type rotavirus strain of non-G1 serotype. Vaccine efficacy (VE) was defined as the percent reduction in the frequency of the relevant outcome variable in vaccinated subjects compared with those subjects who received placebo; Test type: Superiority or Other; p = 1, Fisher Exact; Percent reduction = -97.2, 95% CI 2-sided [-9610.8 to 80.5]

6. Secondary Outcome: Number of Subjects With Severe Rotavirus Gastroenteritis (RVGE) With Non-G1 Serotype
Description: Number of rotavirus gastroenteritis (RVGE) episodes caused by the wild-type rotavirus strain of non-G1 serotype and reported during the efficacy period, were presented by severity, using the Vesikari scale. The assessment of intensity of GE episodes was done using the 20-point Vesikari scale, according to which episodes with scores greater than or equal to (≥) 11 were labeled as severe.
Time Frame: During the study period for the long-term follow-up (i.e. 6 months)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1065 | 525
Subjects | 1 | 0
Statistical Analysis 1: Comparison: Rotarix Group vs Placebo Group; Vaccine efficacy with respect to severe rotavirus gastroenteritis (RVGE) caused by the wild-type rotavirus strain of non-G1 serotype was assessed. Vaccine efficacy (VE) was defined as the percent reduction in the frequency of the relevant outcome variable in vaccinated subjects compared with those subjects who received placebo; Test type: Superiority or Other; p = 1, Fisher Exact; Percent reduction = 0, 95% CI 2-sided [0 to 98.7]

7. Secondary Outcome: Number of Subjects With Severe Gastroenteritis (GE)
Description: Severe GE was defined as a GE episode requiring hospitalization and/or re-hydration therapy in a medical facility.
Time Frame: During the study period for the long-term follow-up (i.e. 6 months)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1065 | 525
Subjects | 15 | 6
Statistical Analysis 1: Comparison: Rotarix Group vs Placebo Group; Vaccine efficacy with respect to severe gastroenteritis (GE) was assessed. Vaccine efficacy (VE) was defined as the percent reduction in the frequency of the relevant outcome variable in vaccinated subjects compared with those subjects who received placebo; Test type: Superiority or Other; p = 0.817, Fisher Exact; Percent reduction = -23.2, 95% CI 2-sided [-287.7 to 54.8]

8. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: An SAE was any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the study period for the long-term follow-up (i.e. 6 months)
Population: The analysis was performed on the Total Cohort, which included all subjects who participated in this follow up study with at least one vaccine administration documented in the primary study.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1082 | 531
Subjects | 4 | 7

9. Secondary Outcome: Number of Subjects Reporting Intussusception (IS)
Description: Intussusception is defined as the telescoping of the intestine.
Time Frame: During the period starting from the end of the second follow-up up to the start of the study (up to 6 months)
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1082 | 531
Subjects | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): during the study period for the long-term follow-up (i.e. 6 months)
Arm/Group | Rotarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 4/1082 | 7/531
Other Adverse Events (participants affected / at risk) | 0/1082 | 0/531
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=1082) | Placebo Group (N=531)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Febrile convulsion (Nervous system disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.